CLINICAL TRIAL: NCT03540134
Title: Convection Enhanced Delivery of Autologous Cerebral Spinal Fluid Improves MRI Visualizations of Basal Ganglion Nuclei During Deep Brain Stimulation Surgery
Brief Title: Convection Enhanced Delivery of CSF in DBS for Parkinson's
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jeff Elias, MD (Other)
Responsible Party: Sponsor-Investigator, Jeff Elias, MD, Professor of Neurological Surgery, University of Virginia
Organization: University of Virginia (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-HSR #20457
Record Dates: First submitted 2018-04-11; First posted 2018-05-30 (Actual); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Parkinson Disease
Keywords: DBS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Intracerebral Infusion of Autologous CSF (Experimental): All subjects will receive the intracerebral infusion of autologous cerebral spinal fluid (CSF) during their deep brain stimulation (DBS) surgery. The DBS surgery will be performed on the targeted nucleus either bilaterally or unilaterally, as previously determined by a multidisciplinary team of neurology, neurosurgery, and neuropsychology. During unilateral DBS surgery, the targeted nucleus will be infused using convection enhanced delivery (CED). The nondominant side will be infused during a bilateral DBS procedure.
  Interventions: Device: Intracerebral Infusion of Autologous Cerebral Spinal Fluid

INTERVENTIONS:
Device: Intracerebral Infusion of Autologous Cerebral Spinal Fluid — Unilateral infusion of 0.5 ml autologous CSF before DBS electrode insertion with MRI monitoring

SUMMARY:
This study will evaluate safety foremost but also the distribution and initial effectiveness of infusion-enhanced, MRI-guided DBS for patients with medication-refractory, Parkinson's disease

DETAILED DESCRIPTION:
This is an open-label, single-arm, pilot study investigating the safety and feasibility of infusion-enhanced, MRI-guided DBS electrode placement. The investigators intend to enroll patients with Parkinson's disease and medically-refractory motor symptoms, who are already planned for MRI-guided DBS electrodes under general anesthesia. The hypothesis of the study is that a convective micro-infusion of autologous CSF will enhance the T2-weighted MRI visualization of the targeted nucleus during image-guided DBS surgery for Parkinson's disease. The investigators will record standard clinical measures of PD at baseline and 6 months following DBS surgery. The study will recruit patients at a rate of approximately one a month and will take less than two years to complete.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, age 30 years and older
2. Subjects with advanced PD who are scheduled for MRI-guided DBS surgery under general anesthesia
3. Subjects who are able and willing to give informed consent and able to attend clinic visits through 6 months
4. The target nucleus, GPi or STN, is visible on MRI so that it can be targeted for the study infusion and then for MRI-guided DBS

Exclusion Criteria:

1. DBS surgery planned in the awake condition with microelectrode recordings and clinical testing
2. Spinal pathology not amenable to lumbar puncture
3. Subjects who have had deep brain stimulation or a prior stereotactic ablation of the basal ganglia
4. Legal incapacity or limited legal capacity as determined by the neuropsychologist
5. Are participating or have participated in another clinical trial in the last 30 days
6. Any illness that in the investigator's opinion preclude participation in this study.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2018-12-18 (Actual); Study Completion 2018-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J Elias, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moosa S, Bond AE, Wang TR, Farzad F, Asthagiri AR, Elias WJ. Stereotactic and Functional Neurosurgery Convection-Enhanced Delivery of Autologous Cerebrospinal Fluid Enhances Basal Ganglia Visualization during MRI-Guided Deep Brain Stimulation Surgery. Stereotact Funct Neurosurg. 2023;101(2):93-100. doi: 10.1159/000528738. Epub 2023 Feb 1. PMID 36724759

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were recruited from the medical clinic.
Period: Overall Study
Arm/Group | Intracerebral Infusion of Autologous CSF
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intracerebral Infusion of Autologous CSF
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.25 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events That Are Related to Treatment
Description: Safety will be determined by an evaluation of the incidence and severity of infusion-related side effects and complications from the first treatment day visit through the 6-month post-treatment time point. All AEs will be reported and categorized by investigators as definitely, probably, possibly, unlikely, or unrelated to the CSF infusion, and/or Parkinson's disease progression. Safety will be assessed by incidence and severity of AEs, including changes in physical examinations and neurological examinations, and the number of discontinuations due to AEs.
Time Frame: 6 months postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Intracerebral Infusion of Autologous CSF
Number analyzed (Participants) | 4
Participants | 2

2. Secondary Outcome: % Change in Un-medicated UPDRS, Motor Subsection (Part III) From Baseline to 6 Months
Description: The efficacy endpoint will be focused on determining the degree of change in motor symptoms as measured from the in-medicated UPDRS, motor subsection (Part III).
Time Frame: 6 months postoperatively in comparison to baseline
Measure: Mean (Standard Deviation); unit: percentage of UPDRS change
Arm/Group | Intracerebral Infusion of Autologous CSF
Number analyzed (Participants) | 4
percentage of UPDRS change | -18.5 (.35)

3. Secondary Outcome: Vd/Vi Ratio
Description: The ratio of the volume of distribution (Vd) immediately following the infusion (Vi) with intraoperative 1.5T MRI, T2-weighted sequences to the volume of the infusion (Vi) will be calculated. Each volume is measured in microliters (uL). The distribution of the infusion by convective properties in a deep brain human nucleus (GPi or STN) will be determined by calculating the Vd/Vi ratio.
Time Frame: Day of Surgery
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Intracerebral Infusion of Autologous CSF
Number analyzed (Participants) | 4
ratio | 2.69 (.17)

4. Secondary Outcome: Baseline Levodopa Medication Equivalents (Milligrams)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: Levodopa medication equivalents (milligr
Arm/Group | Intracerebral Infusion of Autologous CSF
Number analyzed (Participants) | 4
Levodopa medication equivalents (milligr | 1893.3 (246.2)

5. Secondary Outcome: Change in Quality of Life Assessment With PDQ-39 Questionnaire
Description: The PDQ-39 questionnaire includes 39 quality of life questions rated on a scale of 0-4. 0 indicating least frequent (never) and 4 indicating most frequent (always). The mean change in the sum of the PDQ-39 questionnaire is being reported with a overall score of 0 being the best quality of life and a maximum score of 156 being the worst possible quality of life.
Time Frame: 6 months postoperatively in comparison to baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intracerebral Infusion of Autologous CSF
Number analyzed (Participants) | 4
score on a scale | -17.75 (30.8)

ADVERSE EVENTS:
Time Frame: AEs were recorded from the initial consent signing until the 6 month follow up visit.
Description: At each visit patients are examined for any incidence of adverse events.
Arm/Group | Intracerebral Infusion of Autologous CSF
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intracerebral Infusion of Autologous CSF (N=4)
Head pain/Headache (Nervous system disorders) | 2
Word finding difficulty (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT03540134/Prot_SAP_003.pdf